CLINICAL TRIAL: NCT03779477
Title: Effect of "Coping With Stress Program" to Depression and Anxiety Symptoms and Brain Functions in Adolescent at High-Risk for Depression
Brief Title: Effect of Coping With Stress Program to Depression, Anxiety, Brain Functions in Adolescent at High-Risk for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Burcu Özkul, Research Assistant, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 453594
Record Dates: First submitted 2018-12-06; First posted 2018-12-19 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Depression
Keywords: Depression; High-Risk; Adolescent; fMRI
MeSH Terms: conditions — Depression | interventions — Coping Skills

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coping with Stress Course (Experimental): The Coping with Stress Program that consists of 8 sessions will be implemented to the experimental group. 8-10 adolescents will be included in this program. The session frequency will be one session per week. After the completion of 8 sessions, two 90-minute sessions will be carried out each month in the following two months.
  Interventions: Behavioral: Coping with Stress Course
- Control (No Intervention): There will be no intervention in the control group. If the program will be effective, this group will also undergo the Coping with Stress Program after the termination of the study.

INTERVENTIONS:
Behavioral: Coping with Stress Course — The Coping with Stress Program is a group program, which is developed by Clarke and Lewinson (1995) for the prevention of depression in high-risk adolescents. It is based on cognitive-behavioral therapy principles and contains psychoeducation and cognitive-behavioral therapy interventions. There are handbooks available for the group leader of the program and the participating adolescents. In the handbook developed for the group leader, there is detailed information about the objective of each session and the implemented interventions. The adolescents will find lists organized for the fulfillment of the tasks in the handbook prepared for them. The handbooks of the program were translated in Turkish and experts were consulted for their validity.
  Arms: Coping with Stress Course

SUMMARY:
Depression is one of the leading diseases that cause disability, disease burden and threaten public health all over the world. In addition to the economic burdens brought on by depression, it also leads to many individual problems such as deterioration in education, increased psychiatric illnesses in the future, self-harm and suicide. For these reasons, it is important to prevent depression or delay the onset of depression. One of the depression prevention programs, "Coping with Stress Program", is a psychoeducational group program based on cognitive-behavioral therapy and researches shows that the program reduces the rate of diagnosing depression and depressive symptoms in adolescents. Although it is an important mental health problem, studies on adolescent depression are limited in Turkey and existing studies are descriptive and there are no randomized controlled trials. It is believed that this research will encourage studies to prevent depression in Turkey.

The primary aim of this research is to determine the effect of coping with stress program on adolescents' depression and anxiety symptoms, which is applied to adolescents with high risk for depression. The second aim is to examine the changes in brain functions of adolescents participating in the coping with stress program. In the first step, high school students will be screened for depression and adolescents with high levels of depression will be identified. In the second step, randomized controlled experimental design will be used. At the first stage of the study, adolescents with high levels of depression and volunteering to participate in the study will be randomly assigned to the experimental and control groups. After pre-test measurements (determination of depression and anxiety level, functional magnetic resonance imaging (fMRI)), the Coping with Stress Program will be applied to the adolescents in the experimental group. Post-test measures (determination of depression and anxiety level, fMRI) will be performed. The amygdala stimulation test will be used for the fMRI experiment and the data obtained from the fMRI before and after the program will be investigated using the general linear model with Statistical Parametric Mapping (SPM).

DETAILED DESCRIPTION:
Study Type: The study was designed as a randomized controlled trial. Site and Date of the Study: The study will be conducted between October 2018 and January 2020 with the first-year high school students who are registered in the high schools under the governance of Izmir Balcova District National Education Directorate.

Participants: The calculation of the sampling size was based on the Brain Functions outcome. It was recommended that at least 20 subjects should be included in each group for brain imaging studies. Taking into consideration the parametric characteristics of the data, which will be obtained with the scale, the investigators planned to include a total of 60 subjects (30 subjects in each group) in the study. The investigators also planned that 6-10 subjects should be adolescents in each group in experimental group. Experimental group will be evaluated with the help of the Coping with Stress Program.

The sampling process of the study: During the initial phase of the study, adolescents, who will score 19 or more in the Children's Depression Scale, will be determined. The adolescents, who will fulfill the inclusion criteria, will be evaluated by the investigator with the help of the Hamilton Depression Scale. Adolescents, who will have a score equal to or more than 29 will be referred by the investigator to the Outpatient Department of the Children/Adolescent Mental Health at Dokuz Eylül University.

The adolescents, who will fulfill the inclusion criteria, will be informed about the study's objective and methodology during a face-to-face conversation and their families will be informed by phone. The consent form will be handed to the adolescents in order that participants forward it to the parents for signing if they approve the participation of their children in the study. The adolescents, who will accept to participate, will be numbered starting from 1 and they will be randomized in the experimental and control groups with the help of a simple table of randomized numbers (experimental group: 30 subjects; control group: 30 subjects).

In the school, the subjects will undergo pre-test evaluation with Children Depression Scale, The Center for Epidemiological Studies Depression Scale, and Beck's Anxiety Scale after the obtainment of their verbal and written consent. Then 20 adolescents from the experimental group and 20 healthy adolescents will undergo fMRI examination. The individual characteristics of the groups (age, gender, socio-economic status, history of depression in parents) will be compared regarding the significant differences.

Instruments At this phase of the study, the investigators plan to use the following forms, scales, and examinations: Information Questionnaire, Children Depression Scale, The Center for Epidemiological Studies Depression Scale, Beck's Anxiety Scale, Hamilton Depression Rating Scale, 3 Tesla Magnetic Resonance Imaging Device and Functional Magnetic Resonance Imaging (fMRI).

Magnetic Resonance Imaging (MRI) Technique The MRI examinations will be conducted with 3.0 Tesla magnet (Siemens, Erlangen, Germany) using a 12-channel head coil. First, the investigators will obtain structural images with the axial turbo spin echo (TSE) T2-weighted, coronary 3D-SPACE FLAIR (Dark fluid) and 3D-MPRAGE sequences. The obtained images will be immediately examined by the radiologist and interpreted for the presence of a brain anomaly/pathology considered among the inclusion criteria. Subjects without any radio-pathological finding will also be referred to the fMRI examination. The blood oxygen level-dependent (BOLD) technique, which is previously designed in concordance with the task design will be used for the fMRI.

fMRI Task Meta-analyses which are focused on the evaluation of the structural and functional MRI studies of the depression patients, demonstrated anomalies in the amygdala, hippocampus, and subcortical regions. Therefore, the investigators decided to use an fMRI task, which will stimulate these structures. The amygdala stimulation test developed by Hariri, Bookheimer & Mazziotta is widely used in the studies and it was demonstrated that it could strongly and consistently stimulate amygdala.

This test will be performed in a single session and the subjects will be asked to fulfill two different tasks. The first task consists of 3 blocks of cognitive face processing task and the second task consists of 4 blocks of sensorimotor control task. Facial expressions of anger, fear, surprise, and neutral faces from the FACES stimulus set will be used for this purpose (with equal numbers of male and female faces). Face-matching blocks will exhibit three faces, with one on the top and two at the bottom. The expressions will consist of anger, fear, surprise, and neutral outlook. The participant will be asked to match the face on the top with one of the faces at the bottom, which he/she will consider having the same expression. For each face expression (e.g. fear) there will be 6 trials which are equalized for the gender distribution. Each test will last 6 seconds. There will be an interval of 3 seconds between each test (inter-stimulus interval). Each block lasts 54 seconds. In the sensorimotor control blocks, the participant will have 3 geometric shapes (circle, horizontal, and vertical ellipses), one on the top and two at the bottom and will be asked to match the shape on the top with one at the bottom, which he/she will consider as same. Each control block contains 6 different shapes matching and each test lasts 6 seconds. There will be a 3-second inter-stimulus interval between each test. Each block lasts 54 seconds. The blocks will start after a short instruction ("match the shapes" or "match the faces"). The total duration of the fMRI task is 399 seconds. Responses and the response time will be recorded.

Data Collection Implementation 9th grader high school students will be screened during the 2018-2019 school year and the Coping with Stress Program will be implemented in the experimental group, which will consist of 30 students. The demographic data of each student in the experimental and control groups will be collected with a data collection questionnaire before the start of the study (pre-test measurements).

After the pre-test measurements, 20 volunteers from the control group will be scheduled for the fMRI examination. The adolescents and their family will be instructed about the measures, which are to be considered at the examination day and the adolescents will be informed that he/she should not fasten before the examination. On the examination day, the adolescents will be interviewed in the room of the Standardization of Computational Anatomy Techniques fıor Cognitive and Behavioral Sciences (SoCAT) research group in the Ege University, Department of Mental Health, and Psychiatry. During the interview, the adolescents will receive instructions about the fMRI task. During this instruction, which will last approx. 15 minutes, a facial expression set, a shorter version of the set used during the fMRI examination, will be implemented. The adolescents, who have completed the instruction, will be referred to the 3 Tesla MRI unit of the Radiology Department in Ege University and will undergo MRI examination. The fMRI examination will be performed between 10:00-14:00 in weekends, as the unit is overloaded in weekdays. The adolescents will be asked not to move in the MRI device and will be informed that the fMRI process will start just after the structural imaging is completed. The structural imaging will last approx. 5 minutes and will be followed by the fMRI. During the whole process, the investigator Burcu Özkul and the radiology technician will be present in the MRI unit. Healthy adolescents will also undergo fMRI.

The subjects in the experimental group will undergo the Coping with Stress Program. There will be no intervention in the control group; only pre-test, final test and monitoring measurements will be performed. After the completion of the program implemented in the experimental group (final test), all measurements will be repeated in the 3rd, 6th and 12th months in both experimental and control groups. fMRI imaging will be repeated for the subjects in the experimental group in the 2nd month.

Data Analysis The data obtained during the study will be analyzed with the Statistical Package for the Social Sciences (SPSS) v.22 software package. Demographic data will be expressed with descriptive statistics, such as percentage, mean, and standard deviation. The distribution of the continuous data will be analyzed with the Kolmogorov-Smirnov Test and the homogeneity of the groups will be evaluated with Chi-square test. Regarding the repeated comparative measurements performed before the start of the program, they will be evaluated after the instruction, in the 3rd, 6th and 12th months with the variance analysis.

fMRI Analysis: The images in DICOM format will be uploaded in the SPM 12 software and the standard pre-processing will be carried out. This process constitutes of a re-alignment process (aligning of the images in the time sequence in a 3D format), the normalization to the standard space (MNI) and finally the smoothing process. A general linear model (GLM) will be used for the statistical analysis. Therefore, the common and different neural circuits between the groups will be determined. The p-value of 0.05 will be considered as statistically significant for the intergroup comparisons (after the correction according to the multiple comparisons with the family-wise error correction). The minimum cluster threshold will be limited to 5 voxels.

ELIGIBILITY:
Inclusion Criteria:

* Being first-grader high school student
* Being volunteer for participation in the study
* Obtaining the consent of parents' adolescent
* Being literate
* Fluent speaking and understanding of Turkish language
* Scores equal to or higher than 19 in the Children Depression Scale

Exclusion Criteria:

* Previously diagnosed with depression
* Previously diagnosed with a psychiatric disease
* Presence of a diagnosis of bipolar I or schizophrenia in parents
* Usage of psychotropic agents
* Previous participation in a cognitive-behavioral therapy (more than 8 sessions)
* Previous head trauma (with a conscious loss more than 3 minutes)
* Any reason preventing the participant to enter the MRI device (pacemaker, prosthesis, claustrophobia, etc.).
* Scores equal to or higher than 29 in the Hamilton Depression Rating Scale.
* Plow
* Presence of a chronic physical disease

Ages: 14 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 57 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2020-02-03 (Actual); Study Completion 2020-02-15 (Actual)

PRIMARY OUTCOMES:
20 of participants' change from baseline brain functions at 2 months assessed by functional Magnetic Resonans Imaging | Data will be collected before the program starts (pretest) and two months after the end of the program
  Functional magnetic resonance imaging measures brain activity by detecting changes associated with blood flow. The amygdala stimulation test will be used for the functional magnetic resonance imaging experiment and the data obtained from the fMRI analysis with Statistical Parametric Mapping (SPM). Functional Magnetic resonance imaging of the participants will be performed with Siemens 3 Tesla MRI device.

SECONDARY OUTCOMES:
Change from baseline depressive symptoms at 3, 6 and 12 months assessed by Children Depression Inventory | Data will be collected before the program starts (pretest), three months,six months and one-year after the end of the program
  Data will be collected by the Children Depression Inventory. 0-54 points can be taken from the Children Depression Inventory. The higher the score indicates the greater the severity of depression.The cutpoint of the scale is 19 points.
Change from baseline depressive symptoms at 3, 6 and 12 months assessed by Center of Epidemiological Studies Depression Scale | Data will be collected before the program starts (pretest), three months,six months and one-year after the end of the program
  Data will be collected by the Center of Epidemiological Studies Depression Scale. 0 to 60 points can be obtained from the Center for Epidemiological Studies Depression Scale and the higher the score indicates the more depressive symptoms.
Change from baseline anxiety symptoms at 3, 6 and 12 months assessed by Beck Anxiety Inventory | Data will be collected before the program starts (pretest), three months,six months and one-year after the end of the program
  Data will be collected by the Beck Anxiety Inventory. The total score ranges from 0 to 63. As the total scores of the scale increase, the level of anxiety of the person increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylul University, Izmir, Balçova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mumford JA. A power calculation guide for fMRI studies. Soc Cogn Affect Neurosci. 2012 Aug;7(6):738-42. doi: 10.1093/scan/nss059. Epub 2012 May 28. PMID 22641837
- [Background] Simmons JP, Nelson LD, Simonsohn U. False-positive psychology: undisclosed flexibility in data collection and analysis allows presenting anything as significant. Psychol Sci. 2011 Nov;22(11):1359-66. doi: 10.1177/0956797611417632. Epub 2011 Oct 17. PMID 22006061
- [Background] Foland-Ross LC, Hardin MG, Gotlib IH. Neurobiological markers of familial risk for depression. Curr Top Behav Neurosci. 2013;14:181-206. doi: 10.1007/7854_2012_213. PMID 22573472
- [Background] Murray EA, Wise SP, Drevets WC. Localization of dysfunction in major depressive disorder: prefrontal cortex and amygdala. Biol Psychiatry. 2011 Jun 15;69(12):e43-54. doi: 10.1016/j.biopsych.2010.09.041. Epub 2010 Dec 15. PMID 21111403
- [Background] Schmaal L, Veltman DJ, van Erp TG, Samann PG, Frodl T, Jahanshad N, Loehrer E, Tiemeier H, Hofman A, Niessen WJ, Vernooij MW, Ikram MA, Wittfeld K, Grabe HJ, Block A, Hegenscheid K, Volzke H, Hoehn D, Czisch M, Lagopoulos J, Hatton SN, Hickie IB, Goya-Maldonado R, Kramer B, Gruber O, Couvy-Duchesne B, Renteria ME, Strike LT, Mills NT, de Zubicaray GI, McMahon KL, Medland SE, Martin NG, Gillespie NA, Wright MJ, Hall GB, MacQueen GM, Frey EM, Carballedo A, van Velzen LS, van Tol MJ, van der Wee NJ, Veer IM, Walter H, Schnell K, Schramm E, Normann C, Schoepf D, Konrad C, Zurowski B, Nickson T, McIntosh AM, Papmeyer M, Whalley HC, Sussmann JE, Godlewska BR, Cowen PJ, Fischer FH, Rose M, Penninx BW, Thompson PM, Hibar DP. Subcortical brain alterations in major depressive disorder: findings from the ENIGMA Major Depressive Disorder working group. Mol Psychiatry. 2016 Jun;21(6):806-12. doi: 10.1038/mp.2015.69. Epub 2015 Jun 30. PMID 26122586
- [Background] Hariri AR, Bookheimer SY, Mazziotta JC. Modulating emotional responses: effects of a neocortical network on the limbic system. Neuroreport. 2000 Jan 17;11(1):43-8. doi: 10.1097/00001756-200001170-00009. PMID 10683827
- [Background] Baranger DAA, Margolis S, Hariri AR, Bogdan R. An earlier time of scan is associated with greater threat-related amygdala reactivity. Soc Cogn Affect Neurosci. 2017 Aug 1;12(8):1272-1283. doi: 10.1093/scan/nsx057. PMID 28379578